CLINICAL TRIAL: NCT03969524
Title: Superadded Value of Functional MRI Techniques in Evaluation of Malignant Breast Cancers Following Clips Guided Neoadjuvant Chemotherapeutic Series
Brief Title: Functional MRI in Predicting Response to Chemotherapy
Acronym: MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Sabet, Assistant lecturer of Radiology, Assiut University
Other Study IDs: MRI in response assesment
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Patients will undergo magnetic resonance imaging (MRI) at baseline (T0) (before NAC) and after the 2nd cycle of neoadjuvant chemotherapy(T2). Histopathological examination (gold standard) of the surgical specimen will be done for each patient and Compared to the results of MRI.

SUMMARY:
• Address the accuracy of functional MRI techniques to predict response to neoadjuvant chemotherapy given to local advanced breast cancer patients with correlation with pathology thus allowing early chemotherapy regimen modification to increase number of patients achieving pathological complete response or save patients from toxic effects of ineffective chemotherapy.

DETAILED DESCRIPTION:
patient selection:

Selection of patients diagnosed with of biopsy proven breast cancer (BIRAD VI ) :

• Inclusion criteria: patient in different age groups with local advanced breast cancer who are eligible for neoadjuvant chemotherapy and breast conservative surgery and in need for clip placement for tumor localization

Breast cancer (BC) is the second most common cancer in the world and by far the most frequent cancer among women. In Egypt the incidence rate of breast cancer is 29.9/100,000 population in the age group of 30-34 years with the highest population among young women. (1).

Management of breast cancer depends upon its stage. Early stages (stage I) with small sized breast masses undergo breast conservative surgery (BCS) while locally advanced breast masses (stage II and III) may require Preoperative administration of Neoadjuvant chemotherapy (NAC) to decrease the tumor burden allowing for BCS instead of mastectomy with no significant difference in disease-free survival for patients receiving breast conservation in comparison to mastectomy.(2, 3)

Patients who achieve a pathologic complete response (pCR; defined as no residual tumor or a minimal residual tumor on histologic analysis) post NAC demonstrate significantly longer disease-free and overall survival rates(4).

Predicting whether a patient will respond or not to the given chemotherapy would allow an early change in chemotherapy regime or early resort to surgery saving patients from potential toxic effects of chemotherapy and provide a greater chance of achieving a pCR.(5, 6)

Imaging is more accurate than clinical examination in monitoring response to therapy. Different imaging modalities including Digital mammography, ultrasound and MRI have been incorporated in predicting tumoral response to NAC however the MRI has the upper hand due to its higher sensitivity.(3)

Assessing tumoral response to chemotherapy based on observing the regression in the tumor size is widely accepted(7). However, changes in tumor microvasculature, cell density can predate tumoral size change therefore the use of Functional MRI techniques as diffusion-weighted MRI (DWI), MR spectroscopy (MRS) or Dynamic Contrast-Enhanced MRI (DCE) can be used to quantify these early histopathological changes in the tumor.(8)

DCE MRI was reported by multiple studies as the optimal imaging tool to determine disease response, with an accuracy of approximately 91% however there is no established cutoff of enhancement determining partial versus complete response.In three recent studies, the routine use of DWI allowed early differentiation between responders and non-responders by at least a 20% increase in apparent diffusion coefficient, thereby allowing for tailoring of chemotherapy. Also it was reported that the addition of DWI to DCE MRI resulted in improved diagnostic performance in predicting residual disease after chemotherapy.(3) 80% to 90% of patients receiving NAC have a significant response rate of the primary tumor to neoadjuvant chemotherapy. However, this significant response complicates the surgical excision because it is difficult to verify accurate localization of the site of the previous tumor. Therefore the use of a radiopaque marker placed in the tumor bed before administrating chemotherapy has been reported as a safe and inexpensive technique that allows later on for wire guided localization of the tumor bed before surgical resection (9).

In a report on patients who underwent clip placement and preoperative chemotherapy indicated that preoperative wire localization of the tumor bed would have been impossible in 35.7% of patients and difficult in 21.4% of patients without the aid of the clip. Dash et al. concluded that the clip placement was valuable in 57% of patients at the time of preoperative needle localization(10). Edeiken and colleagues reported a similar experience with ultrasound-guided implantation of metallic markers. The markers reportedly were the only remaining evidence of the original tumor site in (47%) of patients.

In a study conducted in M. D. Anderson Cancer Center, Houston, Texas in 2007 aiming to determine whether patients with breast cancer who received breast-conservation therapy after neoadjuvant chemotherapy had improved outcomes if radiopaque clips were placed to mark the primary tumor. The study concluded that the omission of tumor bed clips was associated with a hazard ratio of 3.69 for increased local recurrence compared with patients who did have radiopaque clip placement (P =.083;95% confidence interval , 0.84-16.16).(9)

ELIGIBILITY:
Inclusion Criteria:

* patient in different age groups with local advanced breast cancer who are eligible for neoadjuvant chemotherapy and breast conservative surgery and in need for clip placement for tumor localization

Exclusion Criteria:

* Patient with breast cancer who are not eligible for NAC (pregnant patients, multicentric breast cancer, metastatic breast cancer).
* Patients who have received any prior chemotherapy, radiation therapy or tamoxifen therapy for their current breast cancer
* Patients with any general contraindication to MRI as presence of any paramagnetic substance as pacemakers, or those with claustrophobia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Selection of patients diagnosed with of biopsy proven breast cancer (BIRAD VI ) :
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
correlations coefficient between functional techniques of MRI breast and histology | 3 years
  by appropriate statistical test
changes in the different functional technique's parameters according to the type of response. | 3 years
  by appropriate statistical test

CONTACTS AND LOCATIONS:
Overall Officials: Osama HA El-Sayed, Professor, Study Director — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

REFERENCES:
- [Background] Rieber A, Brambs HJ, Gabelmann A, Heilmann V, Kreienberg R, Kuhn T. Breast MRI for monitoring response of primary breast cancer to neo-adjuvant chemotherapy. Eur Radiol. 2002 Jul;12(7):1711-9. doi: 10.1007/s00330-001-1233-x. Epub 2002 Feb 14. PMID 12111062
- [Background] Taourel P, Pages E, Millet I, Bourgier C, Rouanet P, Jacot W, Crochet P, Azria D. Magnetic resonance imaging in breast cancer management in the context of neo-adjuvant chemotherapy. Crit Rev Oncol Hematol. 2018 Dec;132:51-65. doi: 10.1016/j.critrevonc.2018.09.012. Epub 2018 Sep 25. PMID 30447927